CLINICAL TRIAL: NCT06661174
Title: A Cohort Study on the Efficacy of Bariatric Surgery for Rapidly Progressing Diabetic Nephropathy
Acronym: EBSDKD
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hua Meng, Director of the General Surgery Department & Obesity and Metabolic Disease Center of China-Japan Friendship Hospital, China-Japan Friendship Hospital
Other Study IDs: EBSDKD
Record Dates: First submitted 2024-05-22; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Bariatric Surgeries; Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Surgical group
  Interventions: Procedure: Bariatric surgery; Other: Non-surgical therapy
- Non-surgical group
  Interventions: Other: Non-surgical therapy

INTERVENTIONS:
Procedure: Bariatric surgery — Laparoscopic sleeve gastrectomy or laparoscopic gastric bypass based on β-cell function
  Groups: Surgical group
Other: Non-surgical therapy — Diet management，exercise，metformin，GLP-1 receptor agonists and other drugs which can lose weight.

SUMMARY:
Establish a cohort of diabetic kidney disease(DKD) patients with intensive weight loss treatment to evaluate the impact of intensive weight loss treatment on the renal prognosis of DKD and construct a prediction model for the improvement of renal outcomes after weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old;

  * BMI>25Kg/m2 or abdominal obesity (i.e. waist circumference>90cm for men and>85cm for women);

    * eGFR<30ml/min/1.73m2 or urinary microalbumin≥300mg/g, eGFR<60ml/min/1.73m2.

Exclusion Criteria:

* Patients who are taking glucocorticoids;

  * Combined with tumors; ③Combined with autoimmune diseases; ④Serum albumin<25g/L.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with DKD treated with intensive weight loss or traditional treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Total weight loss | 1st, 3rd, 6th and 12th month after intervention, respectively.

SECONDARY OUTCOMES:
Serum creatinine | 1st, 3rd, 6th and 12th month after intervention, respectively.
Glomerular filtration rate | 1st, 3rd, 6th and 12th month after intervention, respectively.
Fasting blood glucose | 1st, 3rd, 6th and 12th month after intervention, respectively.
Average blood glucose from continuous glucose monitoring | 1st, 3rd, 6th and 12th month after intervention, respectively.
Postprandial 2-hour blood glucose | 1st, 3rd, 6th and 12th month after intervention, respectively.
HbA1c | 1st, 3rd, 6th and 12th month after intervention, respectively.
Waist circumference and hip circumference | 1st, 3rd, 6th and 12th month after intervention, respectively.
Urinary microalbumin and other Urinalysis indexes | 1st, 3rd, 6th and 12th month after intervention, respectively.
Medication status | 1st, 3rd, 6th and 12th month after intervention, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Meng, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China